CLINICAL TRIAL: NCT04966533
Title: Characterize Metzker Pigmentary Disorders
Status: Completed | Type: Observational
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: RECHMPL21_0383
Record Dates: First submitted 2021-07-05; First posted 2021-07-19 (Actual); Last update posted 2021-07-19 (Actual); Status verified 2021-07

CONDITIONS: Pigment Dispersion; Mosaicism
Keywords: Metzker pigmentary disorder

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Metzker pigmentary disorders are frequent cause of consultation in pediatric dermatology. The investigators can describe 4 patterns. They must be differentiated from mosaicisms because they aren't associated with neurologic disorders and don't require any follow up.

ELIGIBILITY:
Inclusion criteria:

* Metzker pigmentary disorder, age between birth and 18 years old

Exclusion criteria:

* None

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children coming at the pediatric dermatology consultation with a Metkzer pigmentary disorder between 2005 and 2021
Sampling Method: Probability Sample
Enrollment: 74 (Actual)
Dates: Start 2005-01-01 (Actual); Primary Completion 2021-01-30 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
Metzker pigmentary disorder pattern | 1 day
  Plume of smoke/ Cloud/Flag/ Linear

SECONDARY OUTCOMES:
Rate of Evolution | 1 day
  Stability/ partial regression/aggravation

CONTACTS AND LOCATIONS:
Overall Officials: Didier BESSIS, PhD, Study Director — University Hospitals of Montpellier
Locations (1):
- Uh Montpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided
NC